CLINICAL TRIAL: NCT04515979
Title: A Phase 2, Open-label, Multicenter Study to Assess the Efficacy and Safety of Vactosertib in Combination with Pembrolizumab As a First-line Treatment for Subjects with PD-L1 Positive Advanced Non-Small Cell Lung Cancer
Brief Title: Vactosertib in Combination with Pembrolizumab for PD-L1 Positive Non-small Cell Lung Cancer (NSCLC) Subjects
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This is because Medpacto decided to modify its development strategy as the business and development environment changed.
Sponsor: MedPacto, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP-VAC-205; MK3475 B37 (Other: Merck)
Record Dates: First submitted 2020-08-11; First posted 2020-08-17 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — vactosertib; BID protein, human; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- vactosertib+Pembrolizumab (Experimental): Vactosertib (5days on and 2days off) Pembrolizumab 200mg Q3Weeks
  Interventions: Drug: Vactosertib 300 mg BID and pembrolizumab 200 mg IV

INTERVENTIONS:
Drug: Vactosertib 300 mg BID and pembrolizumab 200 mg IV — Vactosertib 300 mg orally (PO) BID(5 days on/2days off) and pembrolizumab 200 mg IV (Q3W).
  Other Names: Vactosertib 300 mg BID and keytruda 200 mg IV

SUMMARY:
This is Phase 2, open label, multi-center study to assess safety and efficacy of vactosertib in combination with pembrolizumab as 1st line treatment for subjects with advanced or metastatic, PD-L1 positive, non-small cell lung cancer (NSCLC) who have not previously received systemic therapy for advanced disease and in whom EGFR, ALK, BRAF, ROS1-directed therapy is not indicated.

DETAILED DESCRIPTION:
Approximately 55 NSCLC subjects with PD-L1 tumor proportion score (TPS) ≥ 1% are expected to be enrolled in this study. Subjects' TPS will be determined by PD-L1 IHC 22C3 pharmDx assay performed according to local laboratory regulations prior to study enrollment.

Subjects who received adjuvant or neoadjuvant therapy are permitted onto the study if the therapy was completed at least 12 months prior to the development of metastatic disease.

Eligible subjects will receive:

• Vactosertib 300 mg orally (PO) BID for 5 days with 2 days off period (5 days on/2days off) and pembrolizumab 200 mg IV on Day 1 of every 3-week cycle (Q3W).

ELIGIBILITY:
Inclusion Criteria:

* Have a histologically- or cytologically-documented NSCLC advanced or stage IV lung cancer
* Have confirmation that EGFR, ALK, BRAF, ROS1-directed therapy is not indicated
* Have measurable disease based on RECIST 1.1
* PD-L1 expression is ≥1% as determined by the PD-L1 IHC 22C3 pharmDx assay
* Have a life expectancy of at least 3 months.
* ECOG 0 or 1
* Subjects must be able to swallow tablets and absorb vactosertib.
* Have adequate organ function as indicated by the following laboratory values in

Exclusion Criteria:

* Is currently participating in a study of an investigational agent
* Has received prior systemic cytotoxic chemotherapy for metastatic disease/ antineoplastic biological therapy /Had major surgery / radiation therapy to the lung
* Has received a live vaccine within 30 days prior to the first dose of study drug.
* Is taking prohibited medications
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Had a severe hypersensitivity reaction to treatment with another mAb previously.
* Has severe hypersensitivity to vactosertib and/or any of its excipients

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-08-05 (Actual)

PRIMARY OUTCOMES:
ORR per RECIST 1.1 | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
  ORR in PD-L1≥1% and PD-L1≥50% population per RECIST 1.1 by investigators

CONTACTS AND LOCATIONS:
Overall Officials: Minkyu Heo, Study Director — MedPacto, Inc.
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No